CLINICAL TRIAL: NCT04112160
Title: Prospective Randomized Controlled Trial for Pain Relief After Office Ureteral Stent Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Margaret Pearle, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU 012018-080
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Pain; Urinary Stone; Urinary Calculi
Keywords: stent removal, pain, kidney stones
MeSH Terms: conditions — Pain; Urinary Calculi; Kidney Calculi | interventions — Ketorolac; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Placebo Comparator): normal saline 0.9%
  Interventions: Drug: normal saline
- Ketorolac (Active Comparator): 30 mg of Ketorolac
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — IM injection of either normal saline or Ketorolac
  Other Names: Toradol
  Arms: Ketorolac
Drug: normal saline — normal saline
  Other Names: Placebo
  Arms: control

SUMMARY:
This is a prospective randomized double-blind controlled trial assessing the benefits of intramuscular ketorolac before or immediately after office ureteral stent removal.

DETAILED DESCRIPTION:
Patients who are undergoing cystoscopy with ureteral stent removal at the University of Texas Southwestern Medical Center and have no contraindications to receiving ketorolac will be eligible. Patients will be randomized to receive either a 1 mL injection of ketorolac tromethamine or 1 mL injection of normal saline (0.9%) as the control arm. Ketorolac is a member of the pyrrolo-pyrrole group of non steroid anti inflammatory drugs. The mechanism of action of ketorolac, like that of other NSAIDs, is not completely understood but may be related to prostaglandin synthetase inhibition. The peak analgesic effect occurs within 2-3 hours. If no contraindications exist, ketorolac can be safely given to patients of any age in the 30 mg intramuscular formulation if given as a one time dose according to the package insert.

Normal saline contains 0.9% of Sodium chloride in each mL. Like ketorolac, it is a clear solution and given that there are no major side effects of normal saline it is a good control for our study. It is packaged in a single dose vial that contains 100 mL. It is preservative free and stored at room temperature (20-25°C). Local pain at the injection site may occur, temporarily.

The investigators will specifically look at pain scores before and after stent removal as well as narcotic medication use, telephone calls and/or emergency room visits for pain. Based on the rate of renal colic from our quality improvement project and prior work, the investigators calculated the maximum number of local subjects to be consented for this study to be n=116 (see biostatistics section). The study is expected to last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 to 79 who have undergone a cystoscopy with indwelling double-J ureteral stent placement at Clements University Hospital and are presenting to the office for cystoscopy and stent removal.

Exclusion Criteria:

* eGFR <50
* any active or history of peptic ulcer disease or GI bleeding
* Bleeding disorder, suspected of confirmed cerebrovascular bleeding, hemorrhagic diathesis, or incomplete hemostasis
* Concurrent use of Aspirin 325mg, wafarin, rivaroxaban, apixaban, clopidogrel, or heparin
* Allergic reaction to NSAIDs
* Concurrent use of other NSAIDs within 24 hours
* Pregnancy (ketorolac contraindicated in this population)
* Recent myocardial infarction (MI)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Pearle, MD.PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Johnson BA, Akhtar A, Crivelli J, Steinberg RL, Sasaki J, Street A, Antonelli JA, Pearle MS. Impact of an Enhanced Recovery After Surgery Protocol on Unplanned Patient Encounters in the Early Postoperative Period After Ureteroscopy. J Endourol. 2022 Mar;36(3):298-302. doi: 10.1089/end.2021.0435. Epub 2021 Oct 14. PMID 34569278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Ketorolac
Started | 63 | 62
Completed | 62 | 62
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 46 | 93
  >=65 years | 16 | 16 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57 [47 to 65] | 54 [44 to 66] | 56 [47 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 35 | 31 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 56 | 53 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 62 | 125
Visual Analog Pain (VAS) Pain Scale at the baseline [Median (Inter-Quartile Range); unit: units on a scale] — Scale from 0 (no pain) to 10 (worst pain of one's life), describe how much pain is experienced prior to any intervetion.
  units on a scale | 1 [0 to 3] | 2 [2 to 4] | 2 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unscheduled Return to Clinic or Emergency Room
Description: Any unscheduled in-person clinical encounter secondary to renal colic following ureteral stent removal.
Time Frame: Seven days following ureteral stent removal.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
Participants | 8 | 1

2. Primary Outcome: Median Visual Analog Pain (VAS) Pain Scale Experienced by Participant 24 Hours Following Stent Removal
Description: Perceived pain on a scale of 0-10 (0= no pain, 10= worst pain ever experienced) recorded by phone call 24 hours after stent removal.
Time Frame: Twenty-four hours following ureteral stent removal.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
score on a scale | 2 [0 to 4] | 1 [1 to 4]

3. Primary Outcome: Number of Participants That Experienced an Injection Complication
Description: Determine if there is any infection site pain or reaction. Determine any complications related to administration of the medication.
Time Frame: Within thirty days post injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
Participants | 1 | 1

4. Primary Outcome: Visual Analog Pain (VAS) Pain Scale 7 Days Following Stent Removal.
Description: Perceived pain on a scale of 0-10 (0= no pain, 10= worst pain ever experienced) recorded by phone call 7 days after stent removal.
Time Frame: Seven days following ureteral stent removal.
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-10, 0= no pain)
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
score on a scale (0-10, 0= no pain) | 0 [0 to 1] | 0 [0 to 1]

5. Secondary Outcome: Number of Patients That Required Opioid Medication Following Ureteral Stent Removal
Description: Determine the use of opioid medications in morphine equivalents in the 24 hours following stent removal.
Time Frame: Twenty-four hours following stent removal.
Population: Number of patients that had any opioid use at 24 hours post stent removal.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
Participants | 17 | 17

6. Secondary Outcome: Average Number of Days the Participant Missed Work
Description: Determine amount of missed work or school due to renal colic following ureteral stent removal.
Time Frame: Seven days following stent removal.
Measure: Mean (Standard Deviation); unit: days of missed work
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 62 | 62
days of missed work | 2.3 (3.7) | 2.7 (4.2)

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Control | Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 0/63 | 0/62

LIMITATIONS AND CAVEATS:
There are inherent variations in the size/location of nephrolithiasis, surgical/stent parameters, and patient characteristics that cannot be be defined or controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT04112160/Prot_SAP_ICF_000.pdf